CLINICAL TRIAL: NCT01302067
Title: A 12-Week, Randomized, Double-Blind, Placebo Controlled, Parallel Group, Multicenter Trial In Overactive Bladder Subjects To Confirm The Efficacy Of 8 Mg Fesoterodine Compared To 4 Mg Fesoterodine.
Brief Title: A 12 Week Study to Confirm the Effectiveness of 8mg of Fesoterodine Compared to 4mg of Fesoterodine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A0221095; EIGHT
Record Dates: First submitted 2011-02-18; First posted 2011-02-23 (Estimated); Results first posted 2013-12-24 (Estimated); Last update posted 2014-03-26 (Estimated); Status verified 2014-02

CONDITIONS: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — fesoterodine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Fesoterodine 8mg (Experimental)
  Interventions: Drug: Fesoterodine 8mg
- Fesoterodine 4mg (Experimental)
  Interventions: Drug: Fesoterodine 4mg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fesoterodine 8mg — Oral, 1 tablet per day, 12 weeks duration, 8mg/day
  Arms: Fesoterodine 8mg
Drug: Fesoterodine 4mg — Oral, 1 tablet per day, 12 weeks duration, 4mg/day
  Arms: Fesoterodine 4mg
Drug: Placebo — Oral, 1 tablet per day, 12 weeks duration
  Arms: Placebo

SUMMARY:
This study is designed to confirm if 8mg of fesoterodine is more effective in reducing overactive bladder symptoms than 4mg of fesoterodine. In addition the study is designed to assess if the higher dose reduces the overall effect of overactive bladder on the subject's daily life more than the lower dose. The study also assesses the side effects and safety of the two doses.

ELIGIBILITY:
Inclusion Criteria:

* 6 months overactive bladder symptoms, minimum of 2 urgency urinary incontinence episodes per 24 hours and minimum of 8 micturitions per 24 hours.

Exclusion Criteria:

* Other concurrent and concomitant medication or disease that could put the subjects at additional risk or interfere with the study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2012 (Actual)
Dates: Start 2011-05; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (290):
- United States (162):
  - Urology Centers of Alabama, Birmingham, Alabama
  - Achieve Clinical Research, LLC, Birmingham, Alabama
  - James Gordon McMurray, MD, Huntsville, Alabama
  - Medical Affiliated Research Center, Inc., Huntsville, Alabama
  - Mobile Ob-Gyn, P.C., Mobile, Alabama
  - Montgomery Women's Health Associates, P.C., Montgomery, Alabama
  - Scottsboro Quick Care Clinic, Scottsboro, Alabama
  - Dedicated Clinical Research, Phoenix, Arizona
  - Genova Clinical Research, Tucson, Arizona
  - NEA Baptist Women's Clinic, Jonesboro, Arkansas
  - A Clinic For Women, Little Rock, Arkansas
  - Larry S. Watkins, MD, Little Rock, Arkansas
  - Lynn Institute of the Ozarks, Little Rock, Arkansas
  - May Women's Health Clinic, Little Rock, Arkansas
  - The Office of Dr. Simon Yassear, MD, Carmichael, California
  - Citrus Valley Medical Research, Inc., Glendora, California
  - Grossmont Center for Clinical Research, La Mesa, California
  - Sockolov and Sockolov APC, Sacramento, California
  - Genesis Center for Clinical Research, San Diego, California
  - San Diego Clinical Trials, San Diego, California
  - Clinical Innovations, Inc., Santa Ana, California
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - Urology Associates, PC, Denver, Colorado
  - Genitourinary Surgical Consultants, Denver, Colorado
  - The Women's Clinic of Northern Colorado, Fort Collins, Colorado
  - Women's Health Specialty Care, Farmington, Connecticut
  - South Florida Medical Research, Aventura, Florida
  - Uromedix, Aventura, Florida
  - Meridien Research, Bradenton, Florida
  - Florida Sleep Disorder Center of Brandon, Brandon, Florida
  - PAB Clinical Research, Brandon, Florida
  - Pulmonary Associates of Brandon, Brandon, Florida
  - Meridien Research, Brooksville, Florida
  - Nature Coast Clinical Research, Crystal River, Florida
  - Doctors Medical Center of Walton County, DeFuniak Springs, Florida
  - Avail Clinical Research, LLC, DeLand, Florida
  - SJS Clinical Research, Inc., Destin, Florida
  - Fleming Island Center for Clinical Research, Fleming Island, Florida
  - M & O Clinical Research, LLC, Fort Lauderdale, Florida
  - Florida Urology Physicians, Fort Myers, Florida
  - Urological Research Network, LLC, Hialeah, Florida
  - Nature Coast Clinical Research, Inverness, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Altus Research, Lake Worth, Florida
  - OB-GYN Associates of Mid-Florida, PA, Leesburg, Florida
  - New Horizon Research Center, Miami, Florida
  - Urology Health Team, PLLC, Ocala, Florida
  - Broward Research Group, Pembroke Pines, Florida
  - Clinical Research of Central Florida, Plant City, Florida
  - Southeastern Research Group, Inc., Tallahassee, Florida
  - Meridien Research, Tampa, Florida
  - Advanced OBGYN Associates, West Palm Beach, Florida
  - Clinical Research of Central Florida, Winter Haven, Florida
  - North Fulton Urology, PC, Roswell, Georgia
  - Clinical Research Atlanta, Stockbridge, Georgia
  - North Georgia Clinical Research, Woodstock, Georgia
  - North Georgia Internal Medicine, Woodstock, Georgia
  - Women's Healthcare Associates dba Rosemark WomenCare Specialists, Idaho Falls, Idaho
  - Advanced Clinical Research, Meridian, Idaho
  - Women's Health Practice, Champaign, Illinois
  - Center for Women's Research, Chicago, Illinois
  - Medical and Surgical Specialists, Galesburg, Illinois
  - Clinical Investigation Specialists, Inc., Gurnee, Illinois
  - American Health Network of Indiana, LLC, Avon, Indiana
  - Summit Research Institute, Bloomington, Indiana
  - MediSphere Medical Research Center, LLC, Evansville, Indiana
  - American Health Network of Indiana, LLC, Greenfield, Indiana
  - Metropolitan Urology, Jeffersonville, Indiana
  - Deaconess Clinic Gateway Health Center, Newburgh, Indiana
  - University of Iowa Healthcare, Iowa City, Iowa
  - Health Science Research Center, Pratt, Kansas
  - Women's and Family Care dba GTC Research, Shawnee, Kansas
  - Heartland Research Associates, LLC, Wichita, Kansas
  - Kentucky Medical Research Center, Lexington, Kentucky
  - Commonwealth Biomedical Research, Madisonville, Kentucky
  - Central Kentucky Research Associates, Inc., Mount Sterling, Kentucky
  - Mount Sterling Clinic, Mount Sterling, Kentucky
  - The Office of Dr. Myron I. Murdock, MD, LLC, Greenbelt, Maryland
  - Boston Clinical Trials, Inc., Boston, Massachusetts
  - Beacon Clinical Research, LLC, Brockton, Massachusetts
  - Clinical Research Center of Cape Cod, Inc., Hyannis, Massachusetts
  - Infinity Medical Research, North Dartmouth, Massachusetts
  - DM Clinical Research, Springfield, Massachusetts
  - Clinical Research Institute of Michigan, LLC, Chesterfield, Michigan
  - CRC of Jackson, Jackson, Mississippi
  - Mississippi Urology Clinic, Jackson, Mississippi
  - Midwest Pharmaceutical Research, City of Saint Peters, Missouri
  - Mercy Health Research, St Louis, Missouri
  - Family Health Care Center, Lincoln, Nebraska
  - Women's Clinic of Lincoln, P.C., Lincoln, Nebraska
  - Lincoln Internal Medicine Associates, Lincoln, Nebraska
  - Clinical Research Center of Nevada, Las Vegas, Nevada
  - Virtua Phoenix Ob-Gyn, Moorestown, New Jersey
  - Premier Research, Inc., Trenton, New Jersey
  - United Medical Associates, Binghamton, New York
  - Brooklyn Urology Research Group, Brooklyn, New York
  - Urological Surgeons of Long Island, Garden City, New York
  - Premier Medical Group of the Hudson Valley, Kingston, New York
  - Mid Hudson Medical Research, PLLC, New Windsor, New York
  - Premier Medical Group of the Hudson Valley, Poughkeepsie, New York
  - Upstate Clinical Research Associates, Williamsville, New York
  - Kernodle Clinic, Inc., Burlington, North Carolina
  - American Health Research, Charlotte, North Carolina
  - Carolina Clinical Trials, Concord, North Carolina
  - Carolina Urology Partners, PLLC, Concord, North Carolina
  - Carolinas Research Associates, Harrisburg, North Carolina
  - University Medical Associates, Huntersville, North Carolina
  - Wake Internal Medicine Consultants, Inc., Raleigh, North Carolina
  - Wake Research Associates, LLC, Raleigh, North Carolina
  - PMG Research of Wilmington, LLC, Wilmington, North Carolina
  - Hawthorne Medical Research, Inc. - Hawthorne OB/GYN Associates, Winston-Salem, North Carolina
  - Hawthorne Medical Research, Inc., Winston-Salem, North Carolina
  - Patient Priority Clinical Sites, LLC, Cincinnati, Ohio
  - Rapid Medical Research, Inc., Cleveland, Ohio
  - Columbus Center for Women's Health Research, Columbus, Ohio
  - Columbus Clinical Research, Columbus, Ohio
  - Hometown Urgent Care and Research, Dayton, Ohio
  - HWC Women's Research Center, Englewood, Ohio
  - Ohio Clinical Research, LLC, Willoughby Hills, Ohio
  - The Office of Johnny B. Roy, MD, Edmond, Oklahoma
  - Legacy Clinical Research, LLC, Oklahoma City, Oklahoma
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Institute for Female Pelvic Medicine, Allentown, Pennsylvania
  - Laurel Highlands OB/GYN, Hopwood, Pennsylvania
  - The Clinical Trial Center, LLC, Jenkintown, Pennsylvania
  - Richard Kastelic and Associates, Johnstown, Pennsylvania
  - Clinical Trials Research Services, LLC, Pittsburgh, Pennsylvania
  - Triangle Urological Group, Pittsburgh, Pennsylvania
  - Mount Nittany Medical Center Health Services Inc. dba Mount Nittany Physician Group, State College, Pennsylvania
  - Pish Medical Associates, Uniontown, Pennsylvania
  - Advanced Clinical Concepts, West Reading, Pennsylvania
  - Woman's Clinic Ltd., West Reading, Pennsylvania
  - Coastal Medical, East Greenwich, Rhode Island
  - Safe Harbor Clinical Research, East Providence, Rhode Island
  - Omega Medical Research, Warwick, Rhode Island
  - TLM Medical Services, LLC, Columbia, South Carolina
  - Coastal Carolina Research Center, Mt. Pleasant, South Carolina
  - Southern Urogynecology, West Columbia, South Carolina
  - Internal Medicine and Pediatric Associates of Bristol, PC, Bristol, Tennessee
  - PMG Research of Bristol, LLC, Bristol, Tennessee
  - Adams Patterson Gynocology and Obstetrics, PLLC, Memphis, Tennessee
  - Heartland Medical PC, New Tazewell, Tennessee
  - Austin Center for Clinical Research, Austin, Texas
  - RJE Clinical Research, Dallas, Texas
  - Memorial Clinical Associates dba MCA Research, Houston, Texas
  - ACRC Trials (Administrative/Mailing Site), Plano, Texas
  - North Texas Family Medicine, Plano, Texas
  - Clinical Trials of Texas, Inc., San Antonio, Texas
  - Institute for Women's Health, San Antonio, Texas
  - Seven Oaks Women's Center, San Antonio, Texas
  - Scott and White Healthcare, Temple, Texas
  - Charlottesville Medical Research, Charlottesville, Virginia
  - National Clinical Research - Richmond, Richmond, Virginia
  - Independence Family Medicine, Virginia Beach, Virginia
  - Seattle Urology Research Center, Burien, Washington
  - CAMC Clinical Trials Center, Charleston, West Virginia
  - CAMC Physicians Group, Charleston, West Virginia
  - Charleston Internal Medicine, Inc., Charleston, West Virginia
  - Urologic Surgical Center, Charleston, West Virginia
  - Clinical Investigation Specialists, Inc., Kenosha, Wisconsin
  - Dean Oregon Clinic, Oregon, Wisconsin
  - Allegiance Research Specialists, Wauwatosa, Wisconsin
- Argentina (3):
  - Instituto Urologico Buenos Aires, Buenos Aires
  - Centro de Urología (CDU), Buenos Aires
  - Instituto Medico Especializado (IME), Buenos Aires
- Canada (16):
  - Office of Dr. Peter Pommerville, Victoria, British Columbia
  - Can-Med Clinical Research, Victoria, British Columbia
  - Office of Dr. Nazmuddin Merali, Victoria, British Columbia
  - Can-Med Clinical Research Incorporated, Victoria, British Columbia
  - Pharos Medical Research Ltd., Grand Falls-Windsor, Newfoundland and Labrador
  - Queen Elizabeth Health Sciences Centre, Halifax, Nova Scotia
  - McMaster Institute of Urology, St Joseph's Healthcare Hamilton, Hamilton, Ontario
  - Office of Dr. Bernard Goldfarb, North Bay, Ontario
  - Stanley Flax Medical Professional Corporation, North York, Ontario
  - Urotec, Oshawa, Ontario
  - Toronto Western Hospital, University Health Network, Toronto, Ontario
  - Toronto Urology Clinical Study Group, Toronto, Ontario
  - Urology South Shore Research, Greenfield Park, Quebec
  - UroLaval, Laval, Quebec
  - Ultra-Med Inc., Pointe-Claire, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec
- Chile (2):
  - Clinica Uromed, Santiago, RM
  - Hospital Clinico Universidad de Chile, Santiago, RM
- Colombia (2):
  - Fundacion Centro de Investigacion Clinica CIC, Medellín, Antioquia
  - Solano Y Terront Servicios Medicos Ltda / Unidad Integral de Endocrinologia Uniendo, Bogota, Cundinamarca
- Czechia (7):
  - Urologicka ambulance, Benešov
  - FN a LFUK Hradec Kralove/Urologicka klinika, Hradec Králové
  - Nemocnice Jablonec nad Nisou, Jablonec nad Nisou
  - Fakultni nemocnice v Motole, Prague
  - Urologicka klinika, Praha 1 - Nove Mesto
  - Androgeos spol. s.r.o., Praha 6 - Hradcany
  - Urologicka ambulance, Znojmo
- Denmark (2):
  - Herlev Hospital, Herlev
  - Roskilde sygehus, Gynaekologisk/obstetrisk afdeling, Roskilde
- Al-Azhar University hospital, Cairo, Egypt
- Finland (2):
  - Kouvolan Lääkäriasema, Kouvola
  - Lääkäriasema Cantti Oy, Kuopio
- France (4):
  - Hôpital Edouard Herriot, Lyon
  - CHU de Nantes - Hôtel Dieu, Nantes
  - Hôpital CAREMEAU - Service Urologie/Andrologie, Nîmes
  - Hôpital Tenon - Service d'Urologie, Paris
- Germany (17):
  - Arztpraxis, Alzey
  - Synexus Clinical Research GmbH, Berlin
  - Klinische Forschung Berlin-Buch GmbH, Berlin
  - Synexus Clinical Research GmbH, Bochum
  - Klinische Forschung Dresden GmbH, Dresden
  - Synexus Clinical Research GmbH, Frankfurt am Main
  - Synexus Clinical Research GmbH, Görlitz
  - Clinical Research Hamburg, Hamburg
  - Klinische Forschung Hannover - Mitte GmbH, Hanover
  - Allgemeinmedizin Praktische Aerzte, Karlsruhe
  - Arztpraxis, Lauenburg
  - Synexus Clinical Research GmbH, Leipzig
  - SMO MD GmbH, Magdeburg
  - CRS Clinical Research Service Moenchengladbach GmbH, Mönchengladbach
  - Praxisklinik Urologie Rhein-Ruhr, Muelheim A.d. Ruhr
  - Facharzt fuer Urologie, Reutlingen
  - Klinische Forschung Schwerin GmbH, Schwerin
- Greece (2):
  - University General Hospital of Larisa/ Urology Department, Larissa
  - General Hospital Papageorgiou, Thessaloniki
- Hungary (4):
  - Synexus Magyarorszag Kft., Budapest
  - Jahn Ferenc Del-pesti Korhaz, Urologiai Osztaly, Budapest
  - Debreceni Egyetem Orvos- es Egeszsegtudomanyi Centrum, Urologiai Klinika, Debrecen
  - Josa Andras Oktatokorhaz Egeszsegugyi Szolgaltato Nonprofit Kft., Urologiai osztaly, Nyíregyháza
- Italy (2):
  - Università Magna Graecia di Catanzaro, Catanzaro, Italy
  - Clinica Urologica Centro Trapianti di rene, Foggia
- Lithuania (3):
  - Saules Seimos Medicinos Centras, JSC, Kaunas
  - Mano Seimos Gydytojas, JSC, Klaipėda
  - Seimos Gydytojas, JSC, Vilnius
- Hospital Lomas de San Luis Internacional, San Luis Potosí City, San Luis Potosí, Mexico
- Norway (4):
  - Medi 3 Elverum AS, Elverum
  - Medi 3 Innlandet, Hamar
  - Norsk Helseklinikk AS, c/o Heiaklinikken, Lierskogen
  - Forusakutten AS, Avdeling for oppdragsforskning, Stavanger
- Philippines (3):
  - Perpetual Succour Hospital of Cebu Inc., Cebu City, Cebu
  - Dr. Pablo O. Torre Memorial Hospital, Bacolod City
  - St. Paul's Hospital, Iloilo City
- Poland (4):
  - Klinika Urologii Akademickie Centrum Kliniczne - Szpital Akademii Medycznej w Gdansku, Gdansk
  - NZOZ Centrum Medyczne, Lodz
  - Centrum Urologiczne Sp. z o. o., Mysłowice
  - Nzoz "Nasz Lekarz", Torun
- Russia (3):
  - Non-governmental Healthcare Institution Departmental Clinical Hospital at Barnaul station OAO RZD, Barnaul
  - Rostov State Medical University, Chair of Urology, Rostov-on-Don
  - Research Institute of Obstetrics and Gynaecology D.O. Otta of North-west Department of RAMS, Saint Petersburg
- Slovakia (9):
  - URO CLINIC, s.r.o., Bratislava
  - Ruzinovska poliklinika, a.s., Bratislava
  - Nemocnica s Poliklinikou Svateho Lukasa Galanta, Galanta
  - UROX s.r.o., Piešťany
  - Centrum urologie Povazska Bystrica, s.r.o. urologicka ambulancia, Považská Bystrica
  - Fakultna nemocnica Trencin, Trenčín
  - GYNPOR SK, s.r.o. Urogynekologicka ambulancia, Zvolen
  - UROGYN,s.r.o., Žilina
  - Fakultna nemocnica s poliklinikou Zilina, Žilina
- South Africa (3):
  - Clinical Research Unit, Pretoria, Gauteng
  - Clinix Private Clinic, Vosloorus, Gauteng
  - Mayo Centre, Roodepoort
- South Korea (6):
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University College of Medicine, Department of Urology, Seoul
  - Samsung Medical Center, Seoul
  - Department of Urology, Korea University Anam Hospital, Seoul
  - The Catholic University of Korea Seoul St. Mary's Hospital, Department of Urology, Seoul
  - Asan Medical Center, Department of Urology, Seoul
- Sweden (10):
  - Carema Specialistvard Eslov, Eslöv
  - Hagakliniken, Gothenburg
  - CTC, Sahlgrenska sjukhuset/SU, Gothenburg
  - Probare, Lund
  - Center for Lakemedelsstudier, Malmo
  - Ladulaas kliniska studier, Skene
  - Verksamhet Urologi, Skövde
  - Kvinnokliniken Karolinska Universitetssjukhuset Huddinge, Stockholm
  - S3 Clinical Research Centers, Vällingby
  - Vasterviks sjukhus, Kvinnokliniken, Västervik
- Taiwan (3):
  - Chang Gung Medical Foundation. Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - National Taiwan University Hospital, Department of Urology, Taipei
  - Taipei Veterans General Hospital/Division of Urology, Taipei
- Ukraine (7):
  - RMI "Chernivtsi Regional Clinical Hosp.", Dep. of Urology, BSMU, Chair of Surgery and Urology, Chernivtsi
  - City Hospital #4 of Donetsk, Woman Consultative Department, Donetsk
  - Department of Urology of Donetsk National Medical University at Central City Clinical Hospital #1, Donetsk
  - MTPI "Central City Clinical Hospital #1"/Donetsk National Medical University n.a. M. Gorkiy,, Donetsk
  - Uzhorod City Outpatient Clinic, Prophylaxis Department, Uzhhorod
  - Vinnitsa Regional Clinical Dispensary of Endocrinology, Vinnitsa
  - Urology Dept of Zaporizhzhia Medical Academy of Postgraduate Education, Zaporizhzhia
- United Kingdom (8):
  - Fowey River Practice, Fowey, Cornwall
  - Knowle House Surgery, Plymouth, Devon
  - Ormeau Health Centre, Belfast, Northern Ireland
  - Cambridge University Hospital Trials NHS Trust, Cambridge
  - Southern General Hospital, Glasgow
  - Baillieston Health Centre, Glasgow
  - Sheepcot Medical Centre, Hertfordshire
  - Royal Hallamshire Hospital, Sheffield

REFERENCES:
- [Derived] Stoniute A, Madhuvrata P, Still M, Barron-Millar E, Nabi G, Omar MI. Oral anticholinergic drugs versus placebo or no treatment for managing overactive bladder syndrome in adults. Cochrane Database Syst Rev. 2023 May 9;5(5):CD003781. doi: 10.1002/14651858.CD003781.pub3. PMID 37160401
- [Derived] Wagg AS, Herschorn S, Carlsson M, Fernet M, Oelke M. A plain language summary of the likelihood of symptom relief for patients taking fesoterodine for overactive bladder. J Comp Eff Res. 2022 Sep;11(13):919-925. doi: 10.2217/cer-2022-0041. Epub 2022 Jul 26. PMID 35881009
- [Derived] Chapple C, Schneider T, Haab F, Sun F, Whelan L, Scholfield D, Dragon E, Mangan E. Superiority of fesoterodine 8 mg vs 4 mg in reducing urgency urinary incontinence episodes in patients with overactive bladder: results of the randomised, double-blind, placebo-controlled EIGHT trial. BJU Int. 2014 Sep;114(3):418-26. doi: 10.1111/bju.12678. Epub 2014 Jul 1. PMID 24552358
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0221095&StudyName=A%2012%20week%20study%20to%20confirm%20the%20effectiveness%20of%208mg%20of%20fesoterodine%20compared%20to%204mg%20of%20fesoterodine

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This report presents results of a 12-week study conducted at 241 centers across 27 countries.
Pre-assignment Details: Participants ≥18 years of age with overactive bladder (OAB) symptoms for ≥6 months prior to screening were enrolled. After screening eligible participants were enrolled into the run-in period and received placebo for 2 weeks in a single-blind manner. Participants completed a 3-day bladder diary for 3 days in the week prior to randomization.
Groups:
- Fesoterodine 4 Milligram (mg): Participants received one sustained-release (SR) tablet with 4 mg fesoterodine once daily for 12 weeks.
- Placebo: Participants received one tablet of placebo per day for 12 weeks.
- Fesoterodine 8 mg: Participants received one SR tablet with 4 mg fesoterodine for 1 week, followed by dose escalation to 8 mg once daily for 11 weeks.
Period: Overall Study
Arm/Group | Fesoterodine 4 Milligram (mg) | Placebo | Fesoterodine 8 mg
Started | 790 | 386 | 779
Completed | 712 | 352 | 681
Not Completed | 78 | 34 | 98
Not completed — Death | 0 | 0 | 1
Not completed — Physician Decision | 9 | 5 | 14
Not completed — Lack of Efficacy | 8 | 4 | 2
Not completed — Lost to Follow-up | 9 | 4 | 15
Not completed — Withdrawal by Subject | 13 | 6 | 10
Not completed — Other | 1 | 1 | 3
Not completed — Protocol Violation | 11 | 0 | 8
Not completed — Adverse Event | 27 | 14 | 45

BASELINE CHARACTERISTICS:
Population: The safety analysis set included all participants who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Fesoterodine 4 Milligram (mg) | Placebo | Fesoterodine 8 mg | Total
Number analyzed (Participants) | 790 | 386 | 779 | 1955
Age, Customized [Number; unit: Years]
  <18 | 0 | 0 | 0 | 0
  18 to 44 | 114 | 49 | 99 | 262
  45 to 64 | 380 | 193 | 377 | 950
  >= 65 | 296 | 144 | 303 | 743
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 647 | 316 | 627 | 1590
  Male | 143 | 70 | 152 | 365

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Number of Urgency Urinary Incontinence (UUI) Episodes Per 24 Hours at Week 12.
Description: UUI episodes were defined as those with the Urinary Sensation Scale (USS) rating of 5 in the diary. USS total range 1 to 5: 1. No feeling of urgency, 2. Mild feeling of urgency, 3. Moderate feeling of urgency, 4. Severe feeling of urgency, 5. Unable to hold; leak urine.
Time Frame: Week 12
Population: Full Analysis Set (FAS)included participants receiving 1 dose of assigned study drug and with 1 baseline (BL) or post-BL efficacy assessment. Last observation carried forward (LOCF) was used to impute missing data at Week 12. Participants with baseline UUI >0 per 24 hours & non-missing change from BL to Week 12 were included.
Measure: Least Squares Mean (Standard Error); unit: Episodes per 24 hours
Arm/Group | Fesoterodine 4 Milligram (mg) | Placebo | Fesoterodine 8 mg
Number analyzed (Participants) | 733 | 370 | 718
Episodes per 24 hours | -2.85 (0.09) | -2.22 (0.12) | -3.12 (0.09)
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine 8 mg; Comparisons were done with 2-sided test at 5% significance level. Null hypothesis: mean change from BL in the number of UUI episodes per 24 hours in the 8mg group was same as 4mg group at Week 12. ANCOVA was used to compare 8mg and 4mg arms for numeric change from BL - Week 12. This included terms for treatment, country, centered BL value and centered BL by treatment interaction, in which centered BL (BL - mean BL) was used to ensure that treatment effect was estimated at mean covariate value; Test type: Superiority or Other; p < 0.0001, ANCOVA — Primary comparison was 8 mg VS. 4 mg (closed-testing method). Treatment effect of 8 mg VS. placebo was tested 1st. Treatment difference of 8 mg VS. 4 mg was tested if a statistically significant difference between 8 mg and placebo was shown; Using a closed testing procedure, no adjustments of α-level was needed at each stage of testing. Each was done at the 0.05 significance level; Least squares mean difference = -0.91, 95% CI 2-sided [-1.16 to -0.66], Standard Error of Mean 0.13 — Note- Standard Error of the Mean in the table refers to Standard Error of the Least Squares Mean
Statistical Analysis 2: Comparison: Fesoterodine 4 Milligram (mg) vs Fesoterodine 8 mg; Treatment comparisons were performed with a two-sided test at the 5% significance level; Test type: Superiority or Other; p = 0.0109, ANCOVA — A closed-testing procedure was used for the treatment comparison; Least squares mean difference = -0.27, 95% CI 2-sided [-0.48 to -0.06], Standard Error of Mean 0.11 — Note- Standard Error of the Mean in the table refers to Standard Error of the Least Squares Mean
Statistical Analysis 3: Comparison: Fesoterodine 4 Milligram (mg) vs Placebo; Treatment comparisons were performed with a two-sided test at the 5% significance level; Test type: Superiority or Other; p < 0.0001, ANCOVA — A closed-testing procedure was used for the treatment comparison; Least squares mean difference = -0.64, 95% CI 2-sided [-0.89 to -0.39], Standard Error of Mean 0.13 — Note- Standard Error of the Mean in the table refers to Standard Error of the Least Squares Mean

2. Secondary Outcome: Change From Baseline in Mean Number of Micturitions Per 24 Hours at Week 4.
Description: Micturitions include episodes of voluntary micturition and episodes of UUI.
Time Frame: Week 4
Population: The FAS included all participants who took at least 1 dose of assigned study drug and had at least 1 BL or post-BL efficacy assessment. The analysis included participants with BL Micturition Frequency >0 per 24 hours and non-missing change from BL to Week 4.
Measure: Least Squares Mean (Standard Error); unit: Episodes per 24 hours
Arm/Group | Fesoterodine 4 Milligram (mg) | Placebo | Fesoterodine 8 mg
Number analyzed (Participants) | 715 | 364 | 705
Episodes per 24 hours | -1.95 (0.13) | -1.19 (0.16) | -2.33 (0.13)
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine 8 mg; P-value was based on an ANCOVA model with terms for treatment, pooled country, and centered baseline value; Test type: Superiority or Other; p < 0.0001, ANCOVA — A closed-testing procedure was used for the treatment comparison; Least squares mean difference = -1.13, 95% CI 2-sided [-1.48 to -0.79], Standard Error of Mean 0.18 — Note- Standard Error of the Mean in the table refers to Standard Error of the Least Squares Mean
Statistical Analysis 2: Comparison: Fesoterodine 4 Milligram (mg) vs Fesoterodine 8 mg; P-value was based on an ANCOVA model with terms for treatment, pooled country, and centered baseline value; Test type: Superiority or Other; p = 0.0082, ANCOVA — A closed-testing procedure was used for the treatment comparison; Least squares mean difference = -0.38, 95% CI 2-sided [-0.67 to -0.10], Standard Error of Mean 0.14 — Note- Standard Error of the Mean in the table refers to Standard Error of the Least Squares Mean
Statistical Analysis 3: Comparison: Fesoterodine 4 Milligram (mg) vs Placebo; P-value was based on an ANCOVA model with terms for treatment, pooled country, and centered baseline value; Test type: Superiority or Other; p < 0.0001, ANCOVA — A closed-testing procedure was used for the treatment comparison; Least squares mean difference = -0.75, 95% CI 2-sided [-1.10 to -0.41], Standard Error of Mean 0.18 — Note- Standard Error of the Mean in the table refers to Standard Error of the Least Squares Mean

3. Secondary Outcome: Change From Baseline in Mean Number of Micturitions Per 24 Hours at Week 12.
Description: Micturitions include episodes of voluntary micturition and episodes of UUI.
Time Frame: Week 12
Population: The FAS included all participants who took at least 1 dose of assigned study drug and had at least 1 BL or post-BL efficacy assessment. LOCF was used to impute missing data at Week 12. The analysis included participants with BL Micturition Frequency >0 per 24 hours and non-missing change from BL to Week 12.
Measure: Least Squares Mean (Standard Error); unit: Episodes per 24 hours
Arm/Group | Fesoterodine 4 Milligram (mg) | Placebo | Fesoterodine 8 mg
Number analyzed (Participants) | 733 | 370 | 719
Episodes per 24 hours | -2.45 (0.13) | -1.58 (0.17) | -2.97 (0.13)
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine 8 mg; P-value was based on an ANCOVA model with terms for treatment, pooled country, and centered baseline value; Test type: Superiority or Other; p < 0.0001, ANCOVA — A closed-testing procedure was used for the treatment comparison; Least squares mean difference = -1.40, 95% CI 2-sided [-1.76 to -1.03], Standard Error of Mean 0.19 — Note- Standard Error of the Mean in the table refers to Standard Error of the Least Squares Mean
Statistical Analysis 2: Comparison: Fesoterodine 4 Milligram (mg) vs Fesoterodine 8 mg; P-value was based on an ANCOVA model with terms for treatment, pooled country, and centered baseline value; Test type: Superiority or Other; p = 0.0006, ANCOVA — A closed-testing procedure was used for the treatment comparison; Least squares mean difference = -0.53, 95% CI 2-sided [-0.83 to -0.23], Standard Error of Mean 0.15 — Note- Standard Error of the Mean in the table refers to Standard Error of the Least Squares Mean
Statistical Analysis 3: Comparison: Fesoterodine 4 Milligram (mg) vs Placebo; P-value was based on an ANCOVA model with terms for treatment, pooled country, and centered baseline value; Test type: Superiority or Other; p < 0.0001, ANCOVA — A closed-testing procedure was used for the treatment comparison; Least squares mean difference = -0.87, 95% CI 2-sided [-1.23 to -0.51], Standard Error of Mean 0.19 — Note- Standard Error of the Mean in the table refers to Standard Error of the Least Squares Mean

4. Secondary Outcome: Change From Baseline in Percentage of Micturitions Per 24 Hours at Week 4.
Description: Micturitions include episodes of voluntary micturition and episodes of UUI.
Time Frame: Week 4
Population: as for outcome 2
Measure: Median (Full Range); unit: Episodes per 24 hours
Arm/Group | Fesoterodine 4 Milligram (mg) | Placebo | Fesoterodine 8 mg
Number analyzed (Participants) | 715 | 364 | 705
Episodes per 24 hours | -14.58 [-65.71 to 96.30] | -9.01 [-60.94 to 95.00] | -17.24 [-70.91 to 117.65]
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine 8 mg; P-value was based on a RANKED ANCOVA model with terms for treatment and pooled country with ranked baseline value as a covariate; Test type: Superiority or Other; p < 0.0001, ANCOVA — A closed-testing procedure was used for the treatment comparison; Testing for percent change from baseline was only carried out for given endpoint if corresponding numeric change result was statistically significant
Statistical Analysis 2: Comparison: Fesoterodine 4 Milligram (mg) vs Fesoterodine 8 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0040, ANCOVA — A closed-testing procedure was used for the treatment comparison; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Fesoterodine 4 Milligram (mg) vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — A closed-testing procedure was used for the treatment comparison; [statistical method as in outcome 4, analysis 1]

5. Secondary Outcome: Change From Baseline in Percentage of Micturitions Per 24 Hours at Week 12.
Description: Micturitions include episodes of voluntary micturition and episodes of UUI.
Time Frame: Week 12
Population: as for outcome 3
Measure: Median (Full Range); unit: Episodes per 24 hours
Arm/Group | Fesoterodine 4 Milligram (mg) | Placebo | Fesoterodine 8 mg
Number analyzed (Participants) | 733 | 370 | 719
Episodes per 24 hours | -19.74 [-64.58 to 92.59] | -12.16 [-64.04 to 95.00] | -24.14 [-76.74 to 78.26]
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine 8 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — A closed-testing procedure was used for the treatment comparison; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Fesoterodine 4 Milligram (mg) vs Fesoterodine 8 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — A closed-testing procedure was used for the treatment comparison; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Fesoterodine 4 Milligram (mg) vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — A closed-testing procedure was used for the treatment comparison; [statistical method as in outcome 4, analysis 1]

6. Secondary Outcome: Change From Baseline in Mean Number of UUI Episodes Per 24 Hours at Week 4.
Description: UUI episodes were defined as those with the USS rating of 5 in the diary. USS total range 1 to 5: 1. No feeling of urgency, 2. Mild feeling of urgency, 3. Moderate feeling of urgency, 4. Severe feeling of urgency, 5. Unable to hold; leak urine.
Time Frame: Week 4
Population: The FAS included all participants who took at least 1 dose of assigned study drug and had at least 1 BL or post-BL efficacy assessment. The analysis included participants with BL UUI >0 per 24 hours and non-missing change from BL to Week 4.
Measure: Least Squares Mean (Standard Error); unit: Episodes per 24 hours
Arm/Group | Fesoterodine 4 Milligram (mg) | Placebo | Fesoterodine 8 mg
Number analyzed (Participants) | 715 | 364 | 704
Episodes per 24 hours | -2.55 (0.09) | -1.99 (0.12) | -2.75 (0.09)
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine 8 mg; P-value was based on an ANCOVA model with terms for treatment, pooled country, centered baseline value and centered baseline by treatment interaction; Test type: Superiority or Other; p < 0.0001, ANCOVA — A closed-testing procedure was used for the treatment comparison; Least squares mean difference = -0.76, 95% CI 2-sided [-1.02 to -0.50], Standard Error of Mean 0.13 — Note- Standard Error of the Mean in the table refers to Standard Error of the Least Squares Mean
Statistical Analysis 2: Comparison: Fesoterodine 4 Milligram (mg) vs Fesoterodine 8 mg; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.0662, ANCOVA — A closed-testing procedure was used for the treatment comparison; Least squares mean difference = -0.20, 95% CI 2-sided [-0.41 to 0.01], Standard Error of Mean 0.11 — Note- Standard Error of the Mean in the table refers to Standard Error of the Least Squares Mean
Statistical Analysis 3: Comparison: Fesoterodine 4 Milligram (mg) vs Placebo; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — A closed-testing procedure was used for the treatment comparison; Least squares mean difference = -0.56, 95% CI 2-sided [-0.82 to -0.30], Standard Error of Mean 0.13 — Note- Standard Error of the Mean in the table refers to Standard Error of the Least Squares Mean

7. Secondary Outcome: Change From Baseline in Percentage of UUI Episodes Per 24 Hours at Week 4.
Description: as for outcome 6
Time Frame: Week 4
Population: as for outcome 6
Measure: Median (Full Range); unit: Episodes per 24 hours
Arm/Group | Fesoterodine 4 Milligram (mg) | Placebo | Fesoterodine 8 mg
Number analyzed (Participants) | 715 | 364 | 704
Episodes per 24 hours | -77.78 [-100.00 to 244.44] | -60.50 [-100.00 to 283.33] | -82.48 [-100.00 to 500.00]
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine 8 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — A closed-testing procedure was used for the treatment comparison; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Fesoterodine 4 Milligram (mg) vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — A closed-testing procedure was used for the treatment comparison; [statistical method as in outcome 4, analysis 1]

8. Secondary Outcome: Change From Baseline in Percentage of UUI Episodes Per 24 Hours at Week 12.
Description: as for outcome 6
Time Frame: Week 12
Population: The FAS included all participants who took at least 1 dose of assigned study drug and had at least 1 BL or post-BL efficacy assessment. LOCF was used to impute missing data at Week 12. The analysis included participants with BL UUI >0 per 24 hours and non-missing change from BL to Week 12.
Measure: Median (Full Range); unit: Episodes per 24 hours
Arm/Group | Fesoterodine 4 Milligram (mg) | Placebo | Fesoterodine 8 mg
Number analyzed (Participants) | 733 | 370 | 718
Episodes per 24 hours | -93.75 [-100.00 to 437.50] | -78.89 [-100.00 to 350.00] | -100.00 [-100.00 to 325.00]
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine 8 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — A closed-testing procedure was used for the treatment comparison; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Fesoterodine 4 Milligram (mg) vs Fesoterodine 8 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0006, ANCOVA — A closed-testing procedure was used for the treatment comparison; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Fesoterodine 4 Milligram (mg) vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0001, ANCOVA — A closed-testing procedure was used for the treatment comparison; [statistical method as in outcome 4, analysis 1]

9. Secondary Outcome: Change From Baseline in Mean Number of Micturition-Related Urgency Episodes Per 24 Hours at Week 4.
Description: The mean number of micturition-related urgency episodes per 24 hours was calculated as the total number of micturitions with USS rating of greater than or equal to (>=) 3 divided by the total number of days that diary data was collected at that visit. USS total range 1 to 5: 1. No feeling of urgency, 2. Mild feeling of urgency, 3. Moderate feeling of urgency, 4. Severe feeling of urgency, 5. Unable to hold; leak urine.
Time Frame: Week 4
Population: The FAS included all participants who took at least 1 dose of assigned study drug and had at least 1 BL or post-BL efficacy assessment. The analysis included participants with BL Micturition-related urgency episodes >0 per 24 hours and non-missing change from BL to Week 4.
Measure: Least Squares Mean (Standard Error); unit: Episodes per 24 hours
Arm/Group | Fesoterodine 4 Milligram (mg) | Placebo | Fesoterodine 8 mg
Number analyzed (Participants) | 715 | 364 | 705
Episodes per 24 hours | -2.89 (0.18) | -1.85 (0.23) | -3.40 (0.18)
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine 8 mg; P-value was based on an ANCOVA model with terms for treatment, pooled country, and centered baseline value; Test type: Superiority or Other; p < 0.0001, ANCOVA — A closed-testing procedure was used for the treatment comparison; Least squares mean difference = -1.55, 95% CI 2-sided [-2.04 to -1.06], Standard Error of Mean 0.25 — Note- Standard Error of the Mean in the table refers to Standard Error of the Least Squares Mean
Statistical Analysis 2: Comparison: Fesoterodine 4 Milligram (mg) vs Fesoterodine 8 mg; P-value was based on an ANCOVA model with terms for treatment, pooled country, and centered baseline value; Test type: Superiority or Other; p = 0.0121, ANCOVA — A closed-testing procedure was used for the treatment comparison; Least squares mean difference = -0.52, 95% CI 2-sided [-0.92 to -0.11], Standard Error of Mean 0.21 — Note- Standard Error of the Mean in the table refers to Standard Error of the Least Squares Mean
Statistical Analysis 3: Comparison: Fesoterodine 4 Milligram (mg) vs Placebo; P-value was based on an ANCOVA model with terms for treatment, pooled country, and centered baseline value; Test type: Superiority or Other; p < 0.0001, ANCOVA — A closed-testing procedure was used for the treatment comparison; Least squares mean difference = -1.04, 95% CI 2-sided [-1.52 to -0.55], Standard Error of Mean 0.25 — Note- Standard Error of the Mean in the table refers to Standard Error of the Least Squares Mean

10. Secondary Outcome: Change From Baseline in Mean Number of Micturition-Related Urgency Episodes Per 24 Hours at Week 12.
Description: as for outcome 9
Time Frame: Week 12
Population: The FAS included all participants who took at least 1 dose of assigned study drug and had at least 1 BL or post-BL efficacy assessment. LOCF was used to impute missing data at Week 12. The analysis included participants with BL Micturition-Related Urgency Episodes >0 per 24 hours and non-missing change from BL to Week 12.
Measure: Least Squares Mean (Standard Error); unit: Episodes per 24 hours
Arm/Group | Fesoterodine 4 Milligram (mg) | Placebo | Fesoterodine 8 mg
Number analyzed (Participants) | 733 | 370 | 719
Episodes per 24 hours | -4.23 (0.19) | -2.99 (0.25) | -5.01 (0.19)
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine 8 mg; P-value was based on an ANCOVA model with terms for treatment, pooled country, and centered baseline value; Test type: Superiority or Other; p < 0.0001, ANCOVA — A closed-testing procedure was used for the treatment comparison; Least squares mean difference = -2.02, 95% CI 2-sided [-2.55 to -1.49], Standard Error of Mean 0.27 — Note- Standard Error of the Mean in the table refers to Standard Error of the Least Squares Mean
Statistical Analysis 2: Comparison: Fesoterodine 4 Milligram (mg) vs Fesoterodine 8 mg; P-value was based on an ANCOVA model with terms for treatment, pooled country, and centered baseline value; Test type: Superiority or Other; p = 0.0005, ANCOVA — A closed-testing procedure was used for the treatment comparison; Least squares mean difference = -0.78, 95% CI 2-sided [-1.22 to -0.34], Standard Error of Mean 0.22 — Note- Standard Error of the Mean in the table refers to Standard Error of the Least Squares Mean
Statistical Analysis 3: Comparison: Fesoterodine 4 Milligram (mg) vs Placebo; P-value was based on an ANCOVA model with terms for treatment, pooled country, and centered baseline value; Test type: Superiority or Other; p < 0.0001, ANCOVA — A closed-testing procedure was used for the treatment comparison; Least squares mean difference = -1.24, 95% CI 2-sided [-1.77 to -0.71], Standard Error of Mean 0.27 — Note- Standard Error of the Mean in the table refers to Standard Error of the Least Squares Mean

11. Secondary Outcome: Change From Baseline in Percentage of Micturition-Related Urgency Episodes Per 24 Hours at Week 4.
Description: as for outcome 9
Time Frame: Week 4
Population: as for outcome 9
Measure: Median (Full Range); unit: Participant
Arm/Group | Fesoterodine 4 Milligram (mg) | Placebo | Fesoterodine 8 mg
Number analyzed (Participants) | 715 | 364 | 705
Participant | -23.26 [-100.00 to 280.00] | -14.70 [-100.00 to 716.67] | -27.27 [-100.00 to 150.00]
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine 8 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — A closed-testing procedure was used for the treatment comparison; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Fesoterodine 4 Milligram (mg) vs Fesoterodine 8 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0348, ANCOVA — A closed-testing procedure was used for the treatment comparison; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Fesoterodine 4 Milligram (mg) vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0003, ANCOVA — A closed-testing procedure was used for the treatment comparison; [statistical method as in outcome 4, analysis 1]

12. Secondary Outcome: Change From Baseline in Percentage of Micturition-Related Urgency Episodes Per 24 Hours at Week 12.
Description: as for outcome 9
Time Frame: Week 12
Population: as for outcome 10
Measure: Median (Full Range); unit: Participant
Arm/Group | Fesoterodine 4 Milligram (mg) | Placebo | Fesoterodine 8 mg
Number analyzed (Participants) | 733 | 370 | 719
Participant | -34.88 [-100.00 to 310.00] | -22.73 [-100.00 to 716.67] | -44.29 [-100.00 to 233.33]
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine 8 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — A closed-testing procedure was used for the treatment comparison; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Fesoterodine 4 Milligram (mg) vs Fesoterodine 8 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0002, ANCOVA — A closed-testing procedure was used for the treatment comparison; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Fesoterodine 4 Milligram (mg) vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — A closed-testing procedure was used for the treatment comparison; [statistical method as in outcome 4, analysis 1]

13. Secondary Outcome: Number of Participants With Change From Baseline in Patient Perception of Bladder Condition (PPBC) at Week 12.
Description: PPBC: a self-administered, single-item, questionnaire that asks participants to describe their perception of their bladder-related problems. The PPBC assessment is rated on a 6-point scale: 1=no problems at all, 2=some very minor problems, 3=some minor problems, 4=moderate problems, 5=severe problems, 6=many severe problems. Improvement is defined as negative change from baseline.
Time Frame: Week 12
Population: The FAS included all participants who took at least 1 dose of assigned study drug and had at least 1 BL or post-BL efficacy assessment. The analysis included participants with non-missing change from baseline value at Week 12.
Measure: Number; unit: Participants
Arm/Group | Fesoterodine 4 Milligram (mg) | Placebo | Fesoterodine 8 mg
Number analyzed (Participants) | 700 | 348 | 677
Participants
  Deterioration | 38 | 25 | 27
  No Change | 172 | 122 | 151
  Minor improvement | 210 | 105 | 170
  Major improvement | 280 | 96 | 329
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine 8 mg; Change at Week 12- deterioration, no change, minor improvement and major improvement: Cochran-Mantel-Haenszel (CMH) test with modified ridit scoring controlling for country was used to calculate p-value; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — A closed-testing procedure was used for the treatment comparison
Statistical Analysis 2: Comparison: Fesoterodine 4 Milligram (mg) vs Fesoterodine 8 mg; [analysis description as in outcome 13, analysis 1]; Test type: Superiority or Other; p = 0.0057, Cochran-Mantel-Haenszel — A closed-testing procedure was used for the treatment comparison
Statistical Analysis 3: Comparison: Fesoterodine 4 Milligram (mg) vs Placebo; [analysis description as in outcome 13, analysis 1]; Test type: Superiority or Other; p = 0.0008, Cochran-Mantel-Haenszel — A closed-testing procedure was used for the treatment comparison

14. Secondary Outcome: Number of Participants With Change From Baseline in Urgency Perception Scale (UPS) at Week 12.
Description: UPS: single-item, self-administered validated questionnaire. Participant answered: "Which of the following would typically describe your experience when you have a desire to urinate?" on a 3-point scale, 1=usually not able to hold urine; 2=usually able to hold urine (without leaking) until I reach a toilet if I go to the toilet immediately; 3= usually able to finish what I am doing before going to the toilet (without leaking). Change = observation minus baseline. Results categorized as Deterioration (Negative change); no change (Score change=0); improvement (Positive change).
Time Frame: Week 12
Population: as for outcome 13
Measure: Number; unit: Participants
Arm/Group | Fesoterodine 4 Milligram (mg) | Placebo | Fesoterodine 8 mg
Number analyzed (Participants) | 700 | 348 | 677
Participants
  Deterioration | 37 | 23 | 30
  No change | 361 | 193 | 305
  Improvement | 302 | 132 | 342
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine 8 mg; [analysis description as in outcome 13, analysis 1]; Test type: Superiority or Other; p = 0.0007, Cochran-Mantel-Haenszel — A closed-testing procedure was used for the treatment comparison
Statistical Analysis 2: Comparison: Fesoterodine 4 Milligram (mg) vs Fesoterodine 8 mg; [analysis description as in outcome 13, analysis 1]; Test type: Superiority or Other; p = 0.0091, Cochran-Mantel-Haenszel — A closed-testing procedure was used for the treatment comparison
Statistical Analysis 3: Comparison: Fesoterodine 4 Milligram (mg) vs Placebo; [analysis description as in outcome 13, analysis 1]; Test type: Superiority or Other; p = 0.3901, Cochran-Mantel-Haenszel — A closed-testing procedure was used for the treatment comparison

15. Secondary Outcome: Change From Baseline in Overactive Bladder Questionnaire (OAB-q) Symptom Bother Score at Week 12.
Description: OAB-q: a self-administered, 33-item, questionnaire that assesses how much the participant has been bothered by selected bladder symptoms. Each item rated by participant on Likert scale 1 (not at all) to 6 (a very great deal). Symptom bother score derived as sum of scores for questions 1-8; lowest possible raw score: 8; highest possible score: 48. Data analyzed based on transformation of the score to a 0 to 100 scale [(Actual total raw score - lowest possible value of raw score)/range]*100. Higher scores values indicative of greater symptom bother.
Time Frame: Week 12
Population: as for outcome 13
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Fesoterodine 4 Milligram (mg) | Placebo | Fesoterodine 8 mg
Number analyzed (Participants) | 701 | 347 | 678
Scores on a scale | -30.19 (1.09) | -22.41 (1.43) | -34.88 (1.10)
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine 8 mg; Change at Week 12- ANCOVA model with terms for treatment, pooled country, centered baseline value and centered baseline by treatment interaction was used to calculate p-value; Test type: Superiority or Other; p < 0.0001, ANCOVA — A closed-testing procedure was used for the treatment comparison; Least squares mean difference = -12.47, 95% CI 2-sided [-15.49 to -9.45], Standard Error of Mean 1.54 — Note- Standard Error of the Mean in the table refers to Standard Error of the Least Squares Mean
Statistical Analysis 2: Comparison: Fesoterodine 4 Milligram (mg) vs Fesoterodine 8 mg; [analysis description as in outcome 15, analysis 1]; Test type: Superiority or Other; p = 0.0002, ANCOVA — A closed-testing procedure was used for the treatment comparison; Least squares mean difference = -4.69, 95% CI 2-sided [-7.15 to -2.22], Standard Error of Mean 1.26 — Note- Standard Error of the Mean in the table refers to Standard Error of the Least Squares Mean
Statistical Analysis 3: Comparison: Fesoterodine 4 Milligram (mg) vs Placebo; [analysis description as in outcome 15, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — A closed-testing procedure was used for the treatment comparison; Least squares mean difference = -7.78, 95% CI 2-sided [-10.78 to -4.78], Standard Error of Mean 1.53 — Note- Standard Error of the Mean in the table refers to Standard Error of the Least Squares Mean

16. Secondary Outcome: Change From Baseline in Health Related Quality of Life (HRQL)-Coping Domain and Total Score of Overactive Bladder Questionnaire (OAB-q) at Week 12.
Description: OAB-q: self-administered, 33-item, questionnaire, assesses how much participant has been bothered by selected bladder symptoms. Each item rated on Likert scale 1 (not at all) to 6 (a very great deal). Questions 9 to 33 constitute HRQL, includes domains: concern, coping, sleep, and social function. HRQL domain and total raw score derived as sum of scores. Transformed score range 0 to 100 (Total HRQL or domain) = [(Highest possible raw score-Actual total raw score)/Raw score range]*100. Higher transformed scores indicative of better HRQL.
Time Frame: Week 12
Population: The FAS included all participants who took at least 1 dose of assigned study drug and had at least 1 BL or post-BL efficacy assessment. The analysis included participants with non-missing change from BL value at Week 12.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Fesoterodine 4 Milligram (mg) | Placebo | Fesoterodine 8 mg
Number analyzed (Participants) | 701 | 347 | 677
Scores on a scale | 26.69 (1.18) | 20.91 (1.55) | 31.38 (1.19)
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine 8 mg; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — A closed-testing procedure was used for the treatment comparison; Least squares mean difference = 10.46, 95% CI 2-sided [7.20 to 13.73], Standard Error of Mean 1.67 — Note- Standard Error of the Mean in the table refers to Standard Error of the Least Squares Mean
Statistical Analysis 2: Comparison: Fesoterodine 4 Milligram (mg) vs Fesoterodine 8 mg; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.0006, ANCOVA — A closed-testing procedure was used for the treatment comparison; Least squares mean difference = 4.68, 95% CI 2-sided [2.01 to 7.36], Standard Error of Mean 1.36 — Note- Standard Error of the Mean in the table refers to Standard Error of the Least Squares Mean
Statistical Analysis 3: Comparison: Fesoterodine 4 Milligram (mg) vs Placebo; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.0005, ANCOVA — A closed-testing procedure was used for the treatment comparison; Least squares mean difference = 5.78, 95% CI 2-sided [2.53 to 9.03], Standard Error of Mean 1.66 — Note- Standard Error of the Mean in the table refers to Standard Error of the Least Squares Mean

17. Secondary Outcome: Change From Baseline in Health Related Quality of Life (HRQL)-Concern Domain and Total Score of Overactive Bladder Questionnaire (OAB-q) at Week 12.
Description: as for outcome 16
Time Frame: Week 12
Population: as for outcome 16
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Fesoterodine 4 Milligram (mg) | Placebo | Fesoterodine 8 mg
Number analyzed (Participants) | 701 | 347 | 677
Scores on a scale | 26.82 (1.15) | 20.27 (1.51) | 31.18 (1.16)
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine 8 mg; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — A closed-testing procedure was used for the treatment comparison; Least squares mean difference = 10.91, 95% CI 2-sided [7.73 to 14.09], Standard Error of Mean 1.62 — Note- Standard Error of the Mean in the table refers to Standard Error of the Least Squares Mean
Statistical Analysis 2: Comparison: Fesoterodine 4 Milligram (mg) vs Fesoterodine 8 mg; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.0010, ANCOVA — A closed-testing procedure was used for the treatment comparison; Least squares mean difference = 4.36, 95% CI 2-sided [1.76 to 6.96], Standard Error of Mean 1.33 — Note- Standard Error of the Mean in the table refers to Standard Error of the Least Squares Mean
Statistical Analysis 3: Comparison: Fesoterodine 4 Milligram (mg) vs Placebo; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — A closed-testing procedure was used for the treatment comparison; Least squares mean difference = 6.55, 95% CI 2-sided [3.39 to 9.72], Standard Error of Mean 1.61 — Note- Standard Error of the Mean in the table refers to Standard Error of the Least Squares Mean

18. Secondary Outcome: Change From Baseline in Health Related Quality of Life (HRQL)-Sleep Domain and Total Score of Overactive Bladder Questionnaire (OAB-q) at Week 12.
Description: as for outcome 16
Time Frame: Week 12
Population: as for outcome 16
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Fesoterodine 4 Milligram (mg) | Placebo | Fesoterodine 8 mg
Number analyzed (Participants) | 701 | 347 | 677
Scores on a scale | 21.97 (1.10) | 18.25 (1.45) | 25.71 (1.12)
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine 8 mg; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — A closed-testing procedure was used for the treatment comparison; Least squares mean difference = 7.46, 95% CI 2-sided [4.40 to 10.51], Standard Error of Mean 1.56 — Note- Standard Error of the Mean in the table refers to Standard Error of the Least Squares Mean
Statistical Analysis 2: Comparison: Fesoterodine 4 Milligram (mg) vs Fesoterodine 8 mg; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.0034, ANCOVA — A closed-testing procedure was used for the treatment comparison; Least squares mean difference = 3.74, 95% CI 2-sided [1.24 to 6.23], Standard Error of Mean 1.27 — Note- Standard Error of the Mean in the table refers to Standard Error of the Least Squares Mean
Statistical Analysis 3: Comparison: Fesoterodine 4 Milligram (mg) vs Placebo; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.0164, ANCOVA — A closed-testing procedure was used for the treatment comparison; Least squares mean difference = 3.72, 95% CI 2-sided [0.68 to 6.76], Standard Error of Mean 1.55 — Note- Standard Error of the Mean in the table refers to Standard Error of the Least Squares Mean

19. Secondary Outcome: Change From Baseline in Health Related Quality of Life (HRQL)-Social Interaction Domain and Total Score of Overactive Bladder Questionnaire (OAB-q) at Week 12.
Description: as for outcome 16
Time Frame: Week 12
Population: as for outcome 16
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Fesoterodine 4 Milligram (mg) | Placebo | Fesoterodine 8 mg
Number analyzed (Participants) | 701 | 347 | 677
Scores on a scale | 16.43 (0.89) | 12.61 (1.17) | 20.11 (0.90)
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine 8 mg; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — A closed-testing procedure was used for the treatment comparison; Least squares mean difference = 7.50, 95% CI 2-sided [5.03 to 9.97], Standard Error of Mean 1.26 — Note- Standard Error of the Mean in the table refers to Standard Error of the Least Squares Mean
Statistical Analysis 2: Comparison: Fesoterodine 4 Milligram (mg) vs Fesoterodine 8 mg; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.0004, ANCOVA — A closed-testing procedure was used for the treatment comparison; Least squares mean difference = 3.68, 95% CI 2-sided [1.65 to 5.70], Standard Error of Mean 1.03 — Note- Standard Error of the Mean in the table refers to Standard Error of the Least Squares Mean
Statistical Analysis 3: Comparison: Fesoterodine 4 Milligram (mg) vs Placebo; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.0023, ANCOVA — A closed-testing procedure was used for the treatment comparison; Least squares mean difference = 3.82, 95% CI 2-sided [1.36 to 6.28], Standard Error of Mean 1.25 — Note- Standard Error of the Mean in the table refers to Standard Error of the Least Squares Mean

20. Secondary Outcome: Change From Baseline in Health Related Quality of Life (HRQL)-Total Score of Overactive Bladder Questionnaire (OAB-q) at Week 12.
Description: as for outcome 16
Time Frame: Week 12
Population: as for outcome 16
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Fesoterodine 4 Milligram (mg) | Placebo | Fesoterodine 8 mg
Number analyzed (Participants) | 701 | 347 | 677
Scores on a scale | 23.70 (1.02) | 18.57 (1.33) | 27.94 (1.03)
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine 8 mg; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — A closed-testing procedure was used for the treatment comparison; Least squares mean difference = 9.37, 95% CI 2-sided [6.56 to 12.18], Standard Error of Mean 1.43 — Note- Standard Error of the Mean in the table refers to Standard Error of the Least Squares Mean
Statistical Analysis 2: Comparison: Fesoterodine 4 Milligram (mg) vs Fesoterodine 8 mg; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.0003, ANCOVA — A closed-testing procedure was used for the treatment comparison; Least squares mean difference = 4.23, 95% CI 2-sided [1.93 to 6.53], Standard Error of Mean 1.17 — Note- Standard Error of the Mean in the table refers to Standard Error of the Least Squares Mean
Statistical Analysis 3: Comparison: Fesoterodine 4 Milligram (mg) vs Placebo; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.0003, ANCOVA — A closed-testing procedure was used for the treatment comparison; Least squares mean difference = 5.14, 95% CI 2-sided [2.34 to 7.94], Standard Error of Mean 1.43 — Note- Standard Error of the Mean in the table refers to Standard Error of the Least Squares Mean

21. Secondary Outcome: Percentage of Participants Who Became Dry at Week 4.
Description: Percentage of participants with no UUI episode for the three day diary, the numerator being the number of participants with no UUI at a visit and the denominator the total number of participants with UUI>0 at baseline. UUI episodes defined as those with USS rating of 5 (unable to hold; leak urine) in the diary
Time Frame: Week 4
Population: The FAS included all participants who took at least 1 dose of assigned study drug and had at least 1 BL or post-BL efficacy assessment. The analysis included participants with baseline UUI >0 per 24 hours and non-missing change from baseline to Week 4.
Measure: Number; unit: Percentage of participants
Arm/Group | Fesoterodine 4 Milligram (mg) | Placebo | Fesoterodine 8 mg
Number analyzed (Participants) | 715 | 364 | 704
Percentage of participants | 35.5 | 26.4 | 36.2
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine 8 mg; P-value was obtained from a Cochran-Mantel-Haenszel (CMH) general association test stratified by country; Test type: Superiority or Other; p = 0.0016, Cochran-Mantel-Haenszel — A closed-testing procedure was used for the treatment comparison
Statistical Analysis 2: Comparison: Fesoterodine 4 Milligram (mg) vs Fesoterodine 8 mg; P-value was obtained from a Cochran-Mantel-Haenszel (CMH) general association test stratified by country; Test type: Superiority or Other; p = 0.8121, Cochran-Mantel-Haenszel — A closed-testing procedure was used for the treatment comparison
Statistical Analysis 3: Comparison: Fesoterodine 4 Milligram (mg) vs Placebo; P-value was obtained from a Cochran-Mantel-Haenszel (CMH) general association test stratified by country; Test type: Superiority or Other; p = 0.0015, Cochran-Mantel-Haenszel — A closed-testing procedure was used for the treatment comparison

22. Secondary Outcome: Percentage of Participants Who Became Dry at Week 12.
Description: Percentage of participants with no UUI episode for the three day diary, the numerator being the number of participants with no UUI at a visit and the denominator the total number of participants with UUI >0 at baseline. UUI episodes defined as those with USS rating of 5 (unable to hold; leak urine) in the diary.
Time Frame: Week 12
Population: The FAS included all participants who took at least 1 dose of assigned study drug and had at least 1 BL or post-BL efficacy assessment. Number of participants with Baseline UUI >0 per 24 hours and non-missing change from baseline to Week 12.
Measure: Number; unit: Percentage of participants
Arm/Group | Fesoterodine 4 Milligram (mg) | Placebo | Fesoterodine 8 mg
Number analyzed (Participants) | 733 | 370 | 718
Percentage of participants | 49.2 | 39.5 | 57.8
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine 8 mg; P-value was obtained from a Cochran-Mantel-Haenszel (CMH) general association test stratified by country; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — A closed-testing procedure was used for the treatment comparison
Statistical Analysis 2: Comparison: Fesoterodine 4 Milligram (mg) vs Fesoterodine 8 mg; P-value was obtained from a Cochran-Mantel-Haenszel (CMH) general association test stratified by country; Test type: Superiority or Other; p = 0.0006, Cochran-Mantel-Haenszel — A closed-testing procedure was used for the treatment comparison
Statistical Analysis 3: Comparison: Fesoterodine 4 Milligram (mg) vs Placebo; P-value was obtained from a Cochran-Mantel-Haenszel (CMH) general association test stratified by country; Test type: Superiority or Other; p = 0.0027, Cochran-Mantel-Haenszel — A closed-testing procedure was used for the treatment comparison

ADVERSE EVENTS:
Time Frame: Baseline to 28 days after the last dose of the study drug
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as nonserious in another participant, or one participant may have experienced both a serious and nonserious event during the study.
Arm/Group | Fesoterodine 4 Milligram (mg) | Placebo | Fesoterodine 8 mg
Serious Adverse Events (participants affected / at risk) | 10/790 | 11/386 | 10/779
Other Adverse Events (participants affected / at risk) | 297/790 | 103/386 | 349/779
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fesoterodine 4 Milligram (mg) (N=790) | Placebo (N=386) | Fesoterodine 8 mg (N=779)
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Ulcerative keratitis (Eye disorders) | 1 | 0 | 0
Hemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1 | 0
Chest pain (General disorders) | 1 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0
Herpes simplex ophthalmic (Infections and infestations) | 1 | 0 | 0
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 | 0 | 1
Labyrinthitis (Infections and infestations) | 0 | 1 | 0
Pelvic inflammatory disease (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 0 | 1
Staphylococcal infection (Infections and infestations) | 0 | 1 | 0
Viral infection (Infections and infestations) | 1 | 0 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Post procedural hemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Benign ovarian tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0
Breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Syncope (Nervous system disorders) | 1 | 0 | 0
Endometrial hyperplasia (Reproductive system and breast disorders) | 1 | 0 | 0
Uterine hemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Peripheral artery thrombosis (Vascular disorders) | 1 | 0 | 0
Peripheral ischemia (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fesoterodine 4 Milligram (mg) (N=790) | Placebo (N=386) | Fesoterodine 8 mg (N=779)
Anemia (Blood and lymphatic system disorders) | 1 | 1 | 2
Lymphadenitis (Blood and lymphatic system disorders) | 1 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 2 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 1
Bradycardia (Cardiac disorders) | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 2
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 1
Eustachian tube obstruction (Ear and labyrinth disorders) | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 3 | 1 | 2
Vertigo positional (Ear and labyrinth disorders) | 1 | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 1 | 0
Blepharitis (Eye disorders) | 0 | 1 | 0
Cataract (Eye disorders) | 2 | 0 | 0
Conjunctival irritation (Eye disorders) | 0 | 0 | 1
Dry eye (Eye disorders) | 8 | 3 | 10
Eye allergy (Eye disorders) | 0 | 0 | 1
Eye pain (Eye disorders) | 0 | 0 | 1
Eye swelling (Eye disorders) | 1 | 0 | 0
Glaucoma (Eye disorders) | 0 | 0 | 1
Scintillating scotoma (Eye disorders) | 0 | 1 | 0
Vision blurred (Eye disorders) | 3 | 0 | 4
Visual acuity reduced (Eye disorders) | 1 | 0 | 2
Visual impairment (Eye disorders) | 0 | 0 | 1
Vitreous floaters (Eye disorders) | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 2 | 0 | 4
Abdominal pain (Gastrointestinal disorders) | 5 | 0 | 3
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 1 | 2 | 6
Abnormal faeces (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 12 | 7 | 31
Diarrhoea (Gastrointestinal disorders) | 13 | 4 | 5
Dry mouth (Gastrointestinal disorders) | 102 | 13 | 203
Dyspepsia (Gastrointestinal disorders) | 8 | 0 | 10
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 2
Enteritis (Gastrointestinal disorders) | 0 | 0 | 2
Flatulence (Gastrointestinal disorders) | 1 | 1 | 3
Frequent bowel movements (Gastrointestinal disorders) | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 2 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 5 | 1 | 4
Glossodynia (Gastrointestinal disorders) | 0 | 0 | 2
Hemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1
Hiatus hernia (Gastrointestinal disorders) | 0 | 1 | 0
Lip dry (Gastrointestinal disorders) | 0 | 0 | 2
Nausea (Gastrointestinal disorders) | 11 | 3 | 10
Oesophagitis (Gastrointestinal disorders) | 0 | 1 | 0
Palatal oedema (Gastrointestinal disorders) | 0 | 0 | 1
Peptic ulcer hemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0
Tongue disorder (Gastrointestinal disorders) | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 2 | 1 | 1
Vomiting (Gastrointestinal disorders) | 3 | 0 | 3
Adverse event (General disorders) | 0 | 1 | 0
Asthenia (General disorders) | 0 | 0 | 1
Chest discomfort (General disorders) | 0 | 0 | 2
Chest pain (General disorders) | 1 | 0 | 1
Chills (General disorders) | 0 | 1 | 0
Face oedema (General disorders) | 0 | 0 | 1
Fatigue (General disorders) | 7 | 4 | 7
Inflammation (General disorders) | 0 | 1 | 0
Malaise (General disorders) | 1 | 0 | 0
Nodule (General disorders) | 0 | 0 | 1
Oedema (General disorders) | 0 | 1 | 1
Oedema peripheral (General disorders) | 1 | 0 | 0
Pain (General disorders) | 2 | 0 | 1
Sluggishness (General disorders) | 1 | 0 | 0
Suprapubic pain (General disorders) | 0 | 1 | 0
Thirst (General disorders) | 0 | 1 | 1
Allergic oedema (Immune system disorders) | 0 | 0 | 1
Food allergy (Immune system disorders) | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 1
Seasonal allergy (Immune system disorders) | 1 | 0 | 0
Acute sinusitis (Infections and infestations) | 0 | 0 | 1
Asymptomatic bacteriuria (Infections and infestations) | 2 | 0 | 0
Bacteriuria (Infections and infestations) | 1 | 0 | 0
Bronchitis (Infections and infestations) | 7 | 4 | 5
Cellulitis (Infections and infestations) | 2 | 0 | 3
Cervicitis (Infections and infestations) | 0 | 0 | 1
Cystitis (Infections and infestations) | 6 | 0 | 6
Diverticulitis (Infections and infestations) | 1 | 0 | 0
Ear infection (Infections and infestations) | 1 | 2 | 1
External ear cellulitis (Infections and infestations) | 1 | 0 | 0
Eye infection (Infections and infestations) | 1 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 1
Fungal infection (Infections and infestations) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 2 | 2
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 4
Gastrointestinal infection (Infections and infestations) | 1 | 0 | 0
Gastrointestinal viral infection (Infections and infestations) | 1 | 0 | 0
Gingival infection (Infections and infestations) | 0 | 1 | 0
Herpes simplex (Infections and infestations) | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 1 | 2
Infected bites (Infections and infestations) | 0 | 0 | 1
Influenza (Infections and infestations) | 2 | 1 | 2
Laryngitis (Infections and infestations) | 0 | 0 | 2
Lower respiratory tract infection (Infections and infestations) | 2 | 0 | 2
Lyme disease (Infections and infestations) | 1 | 0 | 0
Mastitis (Infections and infestations) | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 24 | 18 | 17
Oral herpes (Infections and infestations) | 1 | 0 | 1
Pharyngitis (Infections and infestations) | 2 | 0 | 1
Pharyngitis streptococcal (Infections and infestations) | 0 | 0 | 2
Pneumonia (Infections and infestations) | 0 | 0 | 2
Post procedural infection (Infections and infestations) | 0 | 1 | 0
Postoperative wound infection (Infections and infestations) | 0 | 0 | 1
Rash pustular (Infections and infestations) | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Respiratory tract infection viral (Infections and infestations) | 0 | 0 | 1
Rhinitis (Infections and infestations) | 0 | 3 | 0
Sinusitis (Infections and infestations) | 6 | 3 | 5
Subcutaneous abscess (Infections and infestations) | 1 | 0 | 0
Tinea cruris (Infections and infestations) | 1 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 1
Tooth infection (Infections and infestations) | 2 | 0 | 5
Upper respiratory tract infection (Infections and infestations) | 7 | 3 | 5
Urinary tract infection (Infections and infestations) | 16 | 5 | 17
Vaginal infection (Infections and infestations) | 1 | 0 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 1 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0 | 1
Arthropod sting (Injury, poisoning and procedural complications) | 1 | 0 | 0
Burns second degree (Injury, poisoning and procedural complications) | 0 | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 1
Epicondylitis (Injury, poisoning and procedural complications) | 1 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 2 | 0 | 2
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 1 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 3 | 0 | 0
Limb crushing injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Muscle injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Wound (Injury, poisoning and procedural complications) | 0 | 1 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0
Bacterial test positive (Investigations) | 0 | 0 | 1
Biopsy breast (Investigations) | 0 | 1 | 0
Blood glucose increased (Investigations) | 1 | 0 | 0
Blood pressure increased (Investigations) | 2 | 0 | 2
Body temperature increased (Investigations) | 0 | 0 | 1
Glucose urine present (Investigations) | 0 | 1 | 0
Red blood cells urine positive (Investigations) | 1 | 1 | 1
Smear buccal (Investigations) | 1 | 0 | 0
Smear cervix abnormal (Investigations) | 0 | 0 | 1
Weight increased (Investigations) | 1 | 0 | 1
White blood cells urine positive (Investigations) | 1 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 2
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1
Fluid retention (Metabolism and nutrition disorders) | 0 | 1 | 2
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 | 0 | 1
Gout (Metabolism and nutrition disorders) | 1 | 1 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 1
Vitamin B complex deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 1 | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 9 | 0 | 8
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Muscle disorder (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Ageusia (Nervous system disorders) | 0 | 0 | 2
Amnesia (Nervous system disorders) | 1 | 0 | 0
Anosmia (Nervous system disorders) | 0 | 0 | 1
Burning sensation (Nervous system disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 10 | 1 | 2
Dysgeusia (Nervous system disorders) | 5 | 0 | 1
Head discomfort (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 8 | 2 | 12
Hypoaesthesia (Nervous system disorders) | 2 | 1 | 0
Migraine (Nervous system disorders) | 1 | 0 | 1
Neuritis (Nervous system disorders) | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 2 | 0 | 0
Parosmia (Nervous system disorders) | 1 | 0 | 0
Poor quality sleep (Nervous system disorders) | 1 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 1
Radiculitis lumbosacral (Nervous system disorders) | 0 | 0 | 1
Radiculopathy (Nervous system disorders) | 1 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 1
Sinus headache (Nervous system disorders) | 0 | 0 | 1
Somnolence (Nervous system disorders) | 2 | 1 | 1
Vascular encephalopathy (Nervous system disorders) | 0 | 0 | 1
Abnormal dreams (Psychiatric disorders) | 0 | 0 | 1
Aggression (Psychiatric disorders) | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 2
Depression (Psychiatric disorders) | 2 | 0 | 1
Depressive symptom (Psychiatric disorders) | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 2 | 1
Libido decreased (Psychiatric disorders) | 0 | 0 | 1
Loss of libido (Psychiatric disorders) | 0 | 0 | 1
Mood swings (Psychiatric disorders) | 0 | 0 | 1
Performance fear (Psychiatric disorders) | 0 | 0 | 1
Premature ejaculation (Psychiatric disorders) | 0 | 1 | 0
Sleep disorder (Psychiatric disorders) | 0 | 0 | 1
Stress (Psychiatric disorders) | 0 | 0 | 1
Tic (Psychiatric disorders) | 1 | 0 | 0
Bladder pain (Renal and urinary disorders) | 0 | 2 | 1
Bladder prolapse (Renal and urinary disorders) | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 1 | 3 | 5
Enuresis (Renal and urinary disorders) | 1 | 0 | 0
Glycosuria (Renal and urinary disorders) | 0 | 1 | 0
Haematinuria (Renal and urinary disorders) | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0 | 3
Incontinence (Renal and urinary disorders) | 1 | 0 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 2 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1
Nocturia (Renal and urinary disorders) | 0 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 2 | 0
Renal colic (Renal and urinary disorders) | 0 | 1 | 0
Renal cyst (Renal and urinary disorders) | 1 | 0 | 0
Terminal dribbling (Renal and urinary disorders) | 0 | 0 | 1
Urethral pain (Renal and urinary disorders) | 0 | 0 | 1
Urge incontinence (Renal and urinary disorders) | 1 | 0 | 0
Urinary hesitation (Renal and urinary disorders) | 1 | 0 | 2
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 2 | 0 | 2
Urine flow decreased (Renal and urinary disorders) | 0 | 0 | 1
Urine odour abnormal (Renal and urinary disorders) | 0 | 1 | 0
Breast cyst (Reproductive system and breast disorders) | 1 | 0 | 0
Breast mass (Reproductive system and breast disorders) | 0 | 1 | 0
Breast tenderness (Reproductive system and breast disorders) | 1 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 1 | 0
Premenstrual syndrome (Reproductive system and breast disorders) | 0 | 1 | 0
Uterine spasm (Reproductive system and breast disorders) | 0 | 0 | 1
Vaginal discharge (Reproductive system and breast disorders) | 0 | 0 | 2
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 1 | 7
Dry throat (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 4
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 3
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 4
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 2 | 2
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Generalised erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Granuloma annulare (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Intertrigo (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 0 | 3
Rash (Skin and subcutaneous tissue disorders) | 1 | 2 | 3
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Telangiectasia (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Aneurysm repair (Surgical and medical procedures) | 1 | 0 | 0
Cataract operation (Surgical and medical procedures) | 1 | 0 | 0
Haemorrhoid operation (Surgical and medical procedures) | 1 | 0 | 0
Mass excision (Surgical and medical procedures) | 1 | 0 | 0
Mole excision (Surgical and medical procedures) | 0 | 1 | 0
Skin lesion excision (Surgical and medical procedures) | 0 | 1 | 0
Tendon operation (Surgical and medical procedures) | 0 | 1 | 0
Tooth extraction (Surgical and medical procedures) | 0 | 1 | 0
Hot flush (Vascular disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 6 | 3 | 4
Hypotension (Vascular disorders) | 0 | 1 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0 | 0
Tongue dry (Gastrointestinal disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.